CLINICAL TRIAL: NCT01175837
Title: Short-Term Fasting Prior to Systemic Chemotherapy: A Pilot Feasibility Study
Brief Title: Short-Term Fasting Before Chemotherapy in Treating Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MC09C3; NCI-2010-01572 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC09C3 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2010-07-14; First posted 2010-08-05 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Short-term fasting prior to systemic chemotherapy (Experimental): COHORT I: Patients fast 24 hours before day 1 of course 2 of chemotherapy. If fast is well tolerated, patients may escalate fasting by 12 hours for each subsequent course of chemotherapy for up to 3 courses in the absence of unacceptable toxicity.
  COHORT II: Patients fast at the longest fasting regimen found to be safe and tolerable in cohort I before day 1 of each course of course of chemotherapy for up to 4 courses in the absence of unacceptable toxicity.
  Interventions: Other: questionnaire administration; Other: preventative dietary intervention; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: questionnaire administration — Ancillary studies: Pre- and post-fasting side effect questionnaires
Other: preventative dietary intervention — 24, 36, or 48 hour fast prior to chemotherapy
  Other Names: preventative intervention, dietary
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This clinical trial studies short-term fasting before chemotherapy in treating patients with cancer. Fasting before chemotherapy may protect normal cells from the side effects of chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the safety and feasibility of short-term fasting prior to administration of chemotherapy.

SECONDARY OBJECTIVES:

I. Evaluate weight changes in patients who are exposed to short-term fasting prior to chemotherapy.

II. Get a preliminary estimate of the longest feasible fasting period prior to chemotherapy.

III. Evaluate the toxicity profile of systemic chemotherapy treatment in patients who undergo short-term fasting prior to treatment.

IV. Investigate changes in plasma glucose, insulin, Insulin-like growth factor 1 (IGF-1) and IGF-1binding proteins (BP) in patients who undertake short-term fasting.

OUTLINE:

COHORT I: Patients fast 24 hours before day 1 of course 2 of chemotherapy. If fast is well tolerated, patients may escalate fasting by 12 hours for each subsequent course of chemotherapy for up to 3 courses in the absence of unacceptable toxicity.

COHORT II: Patients fast at the longest fasting regimen found to be safe and tolerable in cohort I before day 1 of each course of course of chemotherapy for up to 4 courses in the absence of unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy
* Scheduled to undergo 4 or more cycles of chemotherapy (with or without past chemotherapy treatment); NOTE: Acceptable chemotherapy regimens are those that have all drugs infused on the first day of the chemotherapy cycle over a period =< 8 hours; EXCEPTION: Continuous 5-FU-containing regimens (such as FOLFOX6 and FOLFIRI) are allowed as both the 5-FU bolus as well as the oxaliplatin and irinotecan administration is completed on day 1 of chemotherapy
* Life expectancy of >= 168 days (6 months)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Body mass index (BMI) > 21 kg/m^2
* Weight loss < 5% of body weight in the last 168 days (6 months)
* Adequate renal function (serum creatinine < 1.5 X UNL [upper normal limit] or creatinine clearance > 50 ml/min)
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Provide informed consent
* Ability to complete patient booklet by themselves or with assistance
* Ability and willingness to undergo >= 24-hour fast prior to chemotherapy
* Willingness to be treated at Mayo Clinic Rochester and be available for follow-up
* Patient willing to provide blood samples for correlative research purposes

Exclusion Criteria:

* Any of the following:

  * Pregnant women;
  * Nursing women;
  * Men or women of childbearing potential who are unwilling to employ adequate contraception throughout the study period
* Diabetes mellitus undergoing therapy with insulin or oral agents
* History of low serum glucose (hypoglycemia) or insulinoma
* History of syncope with calorie restriction in the past or other medical comorbidity, which would make fasting potentially dangerous
* On daily medication that may not be safely taken without food; NOTE: Any non-essential medications and herbal/vitamin supplements should be held to minimize stomach upset during fasting; vitamin C use is discouraged
* Active gastric or duodenal peptic ulcer disease
* History of significant cardiac disease, particularly uncompensated congestive heart failure New York Heart Association (NYHA) grade 2 or more or left ventricular ejection fraction (LVEF) < 40% on any prior assessment; NOTE: Assessment of LVEF prior to therapy is not required in the absence of other clinical indicators of heart disease
* Recent history (< 6 months) of cerebrovascular accident or transient ischemic attacks
* History of gout or elevated uric acid level
* Psychiatric conditions that preclude adherence to study protocol
* Serious intercurrent infections or nonmalignant medical illnesses that are uncontrolled or whose control may potentially be jeopardized by the complications of fasting
* Patients receiving parenteral nutrition
* Receiving steroids (except dexamethasone given for nausea prevention before chemotherapy)
* Patients receiving taxotere-containing chemotherapy regimens requiring pre-treatment steroid administration
* Receiving concomitant treatment with insulin-like growth factor (IGF)-receptor blockers or monoclonal antibodies targeting the IGF ligands
* Any of the following (prior to registration):

  * =< 7 days from the time of a minor surgery;
  * =< 21 days from the time of major surgery;
  * =< 21 days from the time of radiation therapy
* Currently enrolled in a concomitant clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-08-13 (Actual); Primary Completion 2013-05-02 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Number of patients hospitalized during fasting period (for reasons that are not attributed to disease or post-operative complications) | Up to 48 hours
Number of patients experiencing greater than or equal to grade 3 adverse event related to the fasting period | Up to 48 hours
Percentage of patients able to achieve designated fasting regimen (i.e., greater than or equal to 50%) | Up to 48 hours

SECONDARY OUTCOMES:
Weight changes in patients who are exposed to short-term fasting prior to chemotherapy | Baseline and 4 months
  Descriptive statistics will be applied to summarize weight changes from baseline for each subsequent course.
Frequency and percentage of the longest feasible fasting period prior to chemotherapy | 4 months
Overall toxicity incidence and profiles by fasting time and patient as per NCI Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | 4 months
  Analyzed by frequency distributions, graphical techniques, and other descriptive measures.
Change in toxicity as assessed by Side Effect Questionnaire and descriptive statistics | Baseline and 4 months
  Assessing symptoms (with 0 being not at all and 10 being as bad as it can be), fasting difficulty (with 0 being very easy and 10 being extremely difficult), and willingness (with 0 being very willing and 10 being not willing at all).
Changes in levels of plasma glucose, insulin, IGF-1 and IGF-1BP in subjects who undertake short-term fasting by descriptive statistics | Baseline and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles Loprinzi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States